CLINICAL TRIAL: NCT04757584
Title: N-of-1 Trials for Deprescribing Beta-blockers in HFpEF
Brief Title: Pilot Deprescribing N-of-1 Trials for Beta-blockers in HFpEF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 19-10020922-01; K76AG064428 (NIH)
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Results first posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure; Heart Failure, Diastolic; Heart Failure With Preserved Ejection Fraction; Cardiac Failure; Heart Disease
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic; Heart Diseases | interventions — Adrenergic beta-Antagonists; Atenolol; Betaxolol; Bisoprolol; Metoprolol; Nebivolol; Nadolol; Propranolol; Acebutolol; Penbutolol; Pindolol; Carvedilol; Labetalol; Sotalol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Beta Blocker ABAB Sequence (Active Comparator): This arm will follow an ABAB sequence. "A" representing ON beta blockers and "B" representing OFF beta blockers. Subjects in this arm will continue their home dose during the initial A period, they will then crossover into Period 2, where dose reduction will begin until they are off of beta blockers. After Period 2, the subjects have the option to decide if they want to be on or off their beta blocker and proceed with the Follow-Up Phase, or continue to Period 3 if they don't feel ready to make that decision to stay on or go off their beta blocker yet. During Period 3, they will restart beta-blockers, gradually up-titrating until reaching their home dose. Finally, during Period 4, we will again conduct a dose reduction until off of beta blockers.
  Interventions: Drug: Beta blockers
- Beta Blocker BABA Sequence (Active Comparator): This arm will follow a BABA sequence. "A" representing ON beta blockers and "B" representing OFF of beta blockers. Subjects in this arm will have their previously prescribed beta blocker dose reduced until they are completely off of beta blockers during Period 1. They will then crossover into Period 2, where uptitration will begin until they are back on their previously prescribed dose of beta blockers. After Period 2, the subjects have the option to decide if they want to be on or off their beta blocker and proceed with the Follow-Up Phase, or continue to Period 3 if they don't feel ready to make that decision to stay on or go off their beta blocker yet. During Period 3, we will again conduct a dose reduction, until the subject is off of beta blockers. Finally, during Period 4, we will up-titrate them back to their home dose of beta blockers.
  Interventions: Drug: Beta blockers

INTERVENTIONS:
Drug: Beta blockers — The intervention is a two-arm crossover withdrawal/ reversal design (On [A] vs Off [B]) with up to 4 periods, each period lasting up to 6 weeks. During the On period (A), subjects will be on their beta blocker. During the Off period (B), their beta blockers will be down-titrated and subsequently discontinued.
  Subjects will be randomized into either ABAB or BABA sequences.
  Other Names: atenolol; betaxolol; bisoprolol; metoprolol; nebivolol; nadolol; propranolol; acebutolol; penbutolol; pindolol; carvedilol; labetalol; sotalol; metoprolol succinate; metoprolol tartrate

SUMMARY:
In this study, we will test the feasibility of N-of-1 trials for deprescribing beta-blockers in patients with Heart Failure with Preserved Ejection Fraction. To achieve this objective we will conduct 16 4-period N-of-1 trials (on vs. off) and subsequently interview participants to better understand feasibility and pragmatism. The N-of-1 trials will be iteratively refined in real-time based on this feedback.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory adults ≥65 years of age with Heart Failure with Preserved Ejection Fraction (HFpEF) according to ACC/AHA guidelines: (signs and symptoms of Heart failure [HF] and ejection fraction [EF] ≥50%)
* Taking Beta blocker

Exclusion Criteria:

* Alternate Causes of HFpEF Syndrome:

  1. Severe valvular disease
  2. Constrictive pericarditis
  3. High output heart failure
  4. Infiltrative cardiomyopathy
* Other compelling indication for beta blocker:

  1. Prior EF < 50%
  2. Hypertrophic cardiomyopathy
  3. Angina symptoms
  4. Acute coronary syndrome, myocardial infarction or coronary artery bypass surgery in prior 3 year
  5. History of ventricular tachycardia
  6. Atrial arrhythmia with hospitalization for rapid ventricular response, prior 1 year
  7. Sinus tachycardia > 100 beats per minute (bpm), atrial arrhythmia with ventricular rate >90 bpm, systolic blood pressure > 160 mmHg
* Clinical instability (N-of-1 trials are appropriate for stable conditions only)

  1. Decompensated HF
  2. Hospitalized in past 30 days
  3. Medication changes or procedures in prior 14 days (to prevent confounding from other interventions), at PI discretion
* Estimated life expectancy <6 months
* Moderate-severe dementia or psychiatric disorder precluding informed consent
* Any condition that, in Principal Investigator's opinion, makes the patient unsuitable for study participation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parag Goyal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Beta Blocker ABAB Sequence: This arm will follow an ABAB sequence. "A" representing ON beta blockers and "B" representing OFF beta blockers. Subjects in this arm will continue their home dose during the initial A period, they will then crossover into Period 2, where dose reduction will begin until they are off of beta blockers. After Period 2, the subjects have the option to decide if they want to be on or off their beta blocker and proceed with the Follow-Up Phase, or continue to Period 3 if they don't feel ready to make that decision to stay on or go off their beta blocker yet. During Period 3, they will restart beta-blockers, gradually up-titrating until reaching their home dose. Finally, during Period 4, we will again conduct a dose reduction until off of beta blockers.
  Beta blockers: The intervention is a two-arm crossover withdrawal/ reversal design (On [A] vs Off [B]) with up to 4 periods, each period lasting up to 6 weeks. During the On period (A), subjects will be on their beta blocker. During the Off period (B), their beta blockers will be down-titrated and subsequently discontinued.
  Subjects will be randomized into either ABAB or BABA sequences.
- Beta Blocker BABA Sequence: This arm will follow a BABA sequence. "A" representing ON beta blockers and "B" representing OFF of beta blockers. Subjects in this arm will have their previously prescribed beta blocker dose reduced until they are completely off of beta blockers during Period 1. They will then crossover into Period 2, where uptitration will begin until they are back on their previously prescribed dose of beta blockers. After Period 2, the subjects have the option to decide if they want to be on or off their beta blocker and proceed with the Follow-Up Phase, or continue to Period 3 if they don't feel ready to make that decision to stay on or go off their beta blocker yet. During Period 3, we will again conduct a dose reduction, until the subject is off of beta blockers. Finally, during Period 4, we will up-titrate them back to their home dose of beta blockers.
  Beta blockers: The intervention is a two-arm crossover withdrawal/ reversal design (On [A] vs Off [B]) with up to 4 periods, each period lasting up to 6 weeks. During the On period (A), subjects will be on their beta blocker. During the Off period (B), their beta blockers will be down-titrated and subsequently discontinued.
  Subjects will be randomized into either ABAB or BABA sequences.
Period: On or Off Beta Blockers Up to 6 Wks
Arm/Group | Beta Blocker ABAB Sequence | Beta Blocker BABA Sequence
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0
Period: Down-titration/Up-titration Up to 6 Wks
Arm/Group | Beta Blocker ABAB Sequence | Beta Blocker BABA Sequence
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0
Period: Up-titration/Down-titration Up to 6 Wks
Arm/Group | Beta Blocker ABAB Sequence | Beta Blocker BABA Sequence
Started | 0 (All 5 subjects on the ABAB Arm chose to complete the intervention phase after the completion of their 2nd period, and move onto the follow-up phase.) | 2 (2 subjects on the BABA Arm chose to complete the intervention phase after the completion of their 2nd period, and move on to the follow-up phase. The remaining 2 subjects on the BABA Arm chose to continue onto a 3rd period.)
Completed | 0 | 2
Not Completed | 0 | 0
Period: Down-titration/Up-Titration Up to 6 Wks
Arm/Group | Beta Blocker ABAB Sequence | Beta Blocker BABA Sequence
Started | 0 | 0 (The remaining 2 subjects on the BABA Arm chose to complete the intervention phase after the completion of their 3rd period, and move on to the follow-up phase.)
Completed | 0 | 0
Not Completed | 0 | 0
Period: Follow-up
Arm/Group | Beta Blocker ABAB Sequence | Beta Blocker BABA Sequence
Started (After each of the subjects complete their intervention phase, they proceed to a follow-up phase, which lasts for 12 months.) | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Beta Blocker ABAB Sequence | Beta Blocker BABA Sequence | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 5 | 4 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Features of a Feasible and Pragmatic Protocol for Deprescribing N-of-1 Trials in Patients With Heart Failure With Preserved Ejection Fraction, as Measured by Qualitative Interview
Description: Qualitative interviews were conducted to assess the feasibility and acceptability of deprescribing N-of-1 trials and participant experiences. Directed content analysis methods were used to develop relevant categories and themes from interview transcript data. Transcripts were coded and analyzed by two team members, consulting additional members to establish consensus where needed. Inter-rater reliability between coders was established.
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Beta Blocker ABAB Sequence | Beta Blocker BABA Sequence
Number analyzed (Participants) | 5 | 4
participants
  Positive attitude towards deprescribing | 4 | 3
  Questions/concerns about deprescribing N-of-1 trials | 2 | 3
  Desire for patient-centered educational materials about deprescribing and N-of-1 trials | 4 | 3
  Desire for short, pragmatic visits | 2 | 2

2. Primary Outcome: Features of a Feasible and Pragmatic Protocol for Deprescribing N-of-1 Trials in Patients With Heart Failure With Preserved Ejection Fraction, as Measured by Qualitative Interview
Description: Qualitative interviews were conducted to assess the feasibility and acceptability of deprescribing N-of-1 trials and participant experiences. Directed content analysis methods were used to develop relevant categories and themes from interview transcript data. Transcripts were coded and analyzed by two team members, consulting additional members to establish consensus where needed. Inter-rater reliability between coders was established. The outcome measure data is the cumulative count of subjects who identified categories and themes from interview transcript data collected during the span of the outcome measure time frame, up to 6 times over 36 weeks.
Time Frame: The maximum amount of time a subject could have been assessed for this outcome measure is 6 times across 36 weeks. This outcome was measured at each end of period visit (weeks 6, 12, 18, 24, 30) and at the end of intervention (weeks 12, 18, 24, 30, or 36)
Measure: Count of Participants; unit: Participants
Arm/Group | Beta Blocker ABAB Sequence | Beta Blocker BABA Sequence
Number analyzed (Participants) | 5 | 4
Participants
  Technologic challenges related to the protocol | 5 | 4
  Desire for study contact that balances safety and pragmatism | 5 | 3
  Feedback on data visualization tool | 5 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were not assessed as part of this study which examined the feasibility and acceptability of deprescribing N-of-1 trials.
Description: Adverse events were not assessed as part of this study which examined the feasibility and acceptability of deprescribing N-of-1 trials. This study record shares a protocol document and subject population with ClinicalTrials.gov record NCT04767061, which is a separate study. Adverse events data were collected and reported for this associated study in ClinicalTrials.gov record NCT04767061.
Arm/Group | Beta Blocker ABAB Sequence | Beta Blocker BABA Sequence
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT04757584/Prot_SAP_001.pdf
  • Informed Consent Form (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT04757584/ICF_002.pdf